CLINICAL TRIAL: NCT00712608
Title: The Evaluation of Cow's Milk Formula - Study B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Carol L. Berseth, MD, Director Medical Affairs North America, Mead Johnson & Company
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 3378-2
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Term Infants
Keywords: Term; Infant; Formula
MeSH Terms: interventions — Infant Formula; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Marketed cow's milk-based formula
  Interventions: Other: Infant formula
- 2 (Experimental): Cow's milk based formula with prebiotics, different level of fatty acids and fat and a different calcium source
  Interventions: Other: Infant formula
- 3 (Experimental): Cow's milk based formula with prebiotic, different level of fatty acids and fat and a different calcium source
  Interventions: Other: Cow's milk infant formula

INTERVENTIONS:
Other: Infant formula — Marketed cow's milk base infant formula 20 kcal/oz
  Other Names: Similar to Enfamil LIPIL with iron
  Arms: 1
Other: Infant formula — cow's milk based infant formula with prebiotics, different level of fatty acids and fat and a different calcium source
  Other Names: No other similar brand names; experimental formula
  Arms: 2
Other: Cow's milk infant formula — Cow's milk based formula with prebiotics, different level of fatty acids and fat and a different calcium source
  Other Names: No other similar brand names; experimental product
  Arms: 3

SUMMARY:
A study to evaluate the growth and development of term infants fed either a marketed cow's milk formula, or an experimental cow's milk formula with prebiotics + a different calcium source + a different level of fatty acids and fat, or an experimental cow's milk formula with prebiotic + a different calcium source + a different level of fatty acids and fat

ELIGIBILITY:
Inclusion Criteria:

* Term infant
* 12-16 days of age
* 37-42 weeks GA

Exclusion Criteria:

* History of chronic disease, congenital malformation
* Feeding difficulties or formula intolerance
* LGA

Ages: 12 Days to 16 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 399 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Rate of weight gain | 106 days

SECONDARY OUTCOMES:
length and head circumference | 106 days

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Berseth, MD, Study Director — Mead Johnson & Company
Locations (22):
- United States (22):
  - Birmingham Pediatric Group, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Dothan, Alabama
  - Central Arkansas Pediatric Clinic, Benton, Arkansas
  - Medical Associates, Fayetteville, Arkansas
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - Palm Beach Clinical Investigation, LLC, West Palm Beach, Florida
  - Welborn Clinic Research, Newburgh, Indiana
  - Woburn Pediatric Associates Research Department, Woburn, Massachusetts
  - Southwestern Medical Clinic, PC, Niles, Michigan
  - Southwestern Medical Clinic, PC, Stevensville, Michigan
  - Aspen Medical Group, Saint Paul, Minnesota
  - The Center for Human Nutrition, Omaha, Nebraska
  - Odyssey Research, Minot, North Dakota
  - Red Lion Pediatrics, Philadelphia, Pennsylvania
  - Primary Physicians Research, Inc, Pittsburgh, Pennsylvania
  - Holston Medical Group, MeadowView Lane, Kingsport, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Retina Foundation of the Southwest, Dallas, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas

REFERENCES:
- [Derived] Ashley C, Johnston WH, Harris CL, Stolz SI, Wampler JL, Berseth CL. Growth and tolerance of infants fed formula supplemented with polydextrose (PDX) and/or galactooligosaccharides (GOS): double-blind, randomized, controlled trial. Nutr J. 2012 Jun 7;11:38. doi: 10.1186/1475-2891-11-38. PMID 22676715